CLINICAL TRIAL: NCT02899975
Title: Interventional Study to Validate a Investigational Fitness and Information Software for Healthy Elderly and Their Informal Caregivers Within the Scope of the EU (European Union) (AAL: Ambient Active Living) Project WeTakeCare
Brief Title: Interventional Validation Study (WeTakeCare-Project)
Acronym: WTCValIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zurich University of Applied Sciences (Other)
Collaborators: Universitat Politècnica de València (Other)
Responsible Party: Principal Investigator, Heidrun Becker, Prof.Dr. phil., Zurich University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ZurichUAS
Record Dates: First submitted 2015-04-14; First posted 2016-09-14 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Prevention Harmful Effects
Keywords: Validation; Information and Fitness Software; Elderly; WeTakeCare
MeSH Terms: interventions — Validation Studies as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Validation Swiss (Other): 20 german talking elderly and the non-professional caregiver will validate a Fitness and Information software
  Interventions: Other: Validation

INTERVENTIONS:
Other: Validation — Validation of fitness and information software for elderly and caregivers. The participants use a Fitness Software for 2-3 months in their own homes. They should use it 3 times a week The aim of this Intervention is to find out if the regularly use of the Software maintains or improves your physical capabilities. The caregivers also use the games and get a lot of Information about supporting the elderly Person in their everyday life
  Other Names: Validation of a fitness and information software

SUMMARY:
The objective of this study is to validate the prototype of the WeTakeCare- system in the real environment (=end users homes) and is embedded in Work-Package 4 (validation and evaluation) with the following main tasks:

T4.1. Definition of methodologies and protocols T4.2. First validation: concept assessment T4.3. Second validation: functional assessment T4.4. Third validation: real environment T4.5. Final check

Within the validation phase III of our project the investigators want to validate the contents of our fitness and information software WeTakeCare with the target group: elderly and their unprofessional caregivers. It runs on the Microsoft Kinect-System, which is authorised in Switzerland, and is in accordance with the prescribing information. The fitness- and information software contains information about strategies and devices which are available in case an older person is not able to perform the everyday movements in a safe and easy way.

Aim of the training and information software is to support elderly to stay independent from others help as long as possible. The mentioned software is not a medical or therapeutical treatment or a medical or therapeutical product. Performed exercises or presented information are highly regarded in the interest of safety and protection of the participants, and serves to prevent physical restrictions or damage .

There is only minimal risk or burden for the participants; the contents of the intervention itself (training of basic motor skills, instruction of strategies and the use of assistive devices to (partly) compensate restrictions in ADL performance, enablement of caregivers) are a standard in rehabilitation of elderly.

The investigators expect the start of the third validation in October 2015.

DETAILED DESCRIPTION:
General study design and justification of design

Type of study: Validation of the prototype of the fitness- and information Software: WeTakeCare (pilot test) in a pre- post design, no comparators

Duration:

* Preparation of the validation study containing: recruiting, pre-screening, assessing, instructing (2-4 month)
* Validation implies the use of the system during expected 3-6 consecutive months, starting soonest in October 2015- (expected) April 2016.

Population to be studied: Healthy elderly (aged 50+) with mild to moderate restrictions in the performance of ADL and their caregivers Number of participants: Involvement of a total of 20 couples in Switzerland. Incorporating 2-5 couples in the first month to allow detection and resolution of any problem.

Study phases

1. "pre testing" of participants eligibility
2. medical check
3. first assessment (first part of baseline measurements)
4. technical installation of the system Installation of the system at the end-users homes will be realized by staff members (See team member list) from the ZHAW.
5. introduction of participants in the practical use of the system (second part of baseline measurements) To guarantee reality of the pilot it will be conducted without altering the environment except if there's environmental elements/factors posing risks to the end-users when performing the exercises/ using the program. The presence of potential risk factors will be controlled by occupational therapists, accompanying the installation of the system. If there's is any risk factor identified (i.e. reduced available space in front of the television screen), OT's (Occupational therapists) will ensure the removal. If a removal is not possible, alternate possibilities will be verified and in case of non-availability this will lead to study exclusion. After installation of the program participants will receive an initial training on functioning by occupational therapists Weekly follow-up controls will also be conducted by OT's (Occupational therapists) (short questionnaire and assessment of improvement of ADL capabilities). These OT's (Occupational therapists) will have received training in the WTC (WeTakeCare-system) use before.
6. Validation phase with a permanent digital log and weekly measurement of…..
7. final assessment (outcome measurements) Methods of minimising bias A description of the measures taken to minimize/avoid bias, including: Randomization, Blinding.

Within the pretesting phase possible participants are screened to validate the cognitive status as well as the physical condition to include only elderly and caregivers which have a benefit from participation.

STUDY INTERVENTION (SPIRIT #11) 8.1 Identity of Investigational Products (treatment / medical device) (ICH/E6 6.2.1, 6.4.2, 6.4.4; AGEK Checklist 2, item 3) Enrolled participants will get the technical appliances and support with the installation of the gadgets. (Kinect I (Microsoft-Kinect) and if necessary an appropriate Laptop) Occupational therapists will give a comprehensive instruction to the system, which also includes clarification of safety precautions.

The participants are free to use the system within their everyday life whenever they want.(Alone or together with their caregivers.)

ELIGIBILITY:
Inclusion Criteria:

* Elderly
* Healthy elderly with mild to moderate restrictions in performance of ADL, support from an informal caregiver
* aged > 50 years
* living in the German-speaking part of Switzerland
* with self-perceived reduced abilities in the performance of ADL and help from an informal caregiver Caregivers
* aged > 18 years
* expenditure of care > i.e. 1-2 times/week; > 1-2 hrs/week,…

Elderly and caregivers

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Good knowledge of German language
* Availability of internet connection

Exclusion Criteria:

* Elderly and caregivers
* presence of environmental risk factors inhibiting the safe accomplishment of the study

Elderly

* Medical restrictions or instability such as

  * History of epilepsy
  * Severe cardiovascular disorders
  * Severe neurological disorders
  * Surgery less than 3 months ago
  * Recent fractures (< 6 weeks ago and/or instable)
  * moderate to severe depression
  * non- correctible hearing and/or visual impairment
  * progressive or terminal illness
  * cognitive restrictions (MMSE score < 24)
* high risk of falling
* Severe restrictions in ADL performance
* living in a care facility
* receiving professional care

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Measuring a change with the assessment "Performance Quality Rating Scale" (PQRS) | Measured in Baseline and Endpoint after 3 month
  Measures the completeness and Quality of performing different daily tasks. We will use this assessment two times to measure a change after the Intervention.

SECONDARY OUTCOMES:
Measuring a change with the assessment "EQ 5D" (assessment from EuroQol-Group (Researcher Network) 5D (=fifth Version) | Measured in Baseline and Endpoint after 3 month
  Question about Quality of life. We will use this assessment two times to measure a change after the intervention
Measuring a change with the assessment "Burden Scale of Family Caregivers (only caregivers)" | Measured in Baseline and Endpoint after 3 month
  Question about stressing or difficult Situation concerning the caregiving.We will use this assessment two times to measure a change after the intervention
Measuring a change with the assessment "SIMPLIT" (Quality Label) | Measured in Baseline and Endpoint after 3 month
  Question about usability of the prototyp. We will use this assessment two times to measure in elderly become familiar with the System while using it. SIMPLIT is a quality label that guarantees that products have been developed with a design aimed at elderly People.
Measuring a change with the assessment "Senior Fitness Test" | Measured in Baseline and Endpoint after 3 month
  Measures endurance, strength, and other physiological abilities of People 60+. We will use this assessment two times to measure a change after the intervention.
Measuring a change with the assessment "Berg Balance Scale" | Measured in Baseline and Endpoint after 3 month
  Measures Balance capabilities. We will use this assessment two times to measure a change after the Intervention
Measuring a change with the assessment "ICON FES" (Iconographical Falls Efficacy Scale) | Measured in Baseline and Endpoint after 3 month
  Image-based assessment to evaluate fear of falling. We will use this assessment two times to measure a change after the Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rakel Poveda, Prof, Principal Investigator — Universitat Politècnica de València

IPD SHARING:
Plan to Share IPD: No